CLINICAL TRIAL: NCT07131319
Title: Spatially Fractionated Radiotherapy (SFRT) Synchronized With Tislelizumab Plus Platinum-based Dual-agent Chemotherapy for Induction Treatment of Initially Unresectable Stage Ⅲ Non-small Cell Lung Cancer: A Clinical Study
Brief Title: SFRT+Tislelizumab+Platinum Chemotherapy for Unresectable Stage III NSCLC
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2025-026
Record Dates: First submitted 2025-04-25; First posted 2025-08-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Carboplatin; Pemetrexed; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SFRT concurrent with tislelizumab and platinum - based doublet chemotherapy (Experimental): SFRT concurrent with immunochemotherapy is given q3w for 3 cycles. Here are details:
  Radiotherapy: Select several 1 - cm - diameter spherical areas in the primary tumor's hypoxic region, 1.5 - 2 cm apart. Each area receives a single 12 - Gy high - dose radiotherapy, precisely targeting the hypoxic part to enhance the effect.
  Chemotherapy & Immunotherapy: 1 - 3 days after radiotherapy, combine 200 mg of tislelizumab with platinum - based doublet chemotherapy. NSCLC chemo - drug combos vary by pathology. For adenocarcinoma, use pemetrexed (500 mg/m² d1) + carboplatin (AUC 5, d1). For other types, use albumin - bound paclitaxel (100 mg/m² d1,8) + carboplatin (AUC 5, d1).
  Interventions: Other: Spatially Fractionated Radiotherapy (SFRT); Drug: Tislelizumab, Carboplatin, Pemetrexed; Drug: Tislelizumab, paclitaxel, Carboplatin

INTERVENTIONS:
Other: Spatially Fractionated Radiotherapy (SFRT) — Several spherical volumes (with a diameter of 1 cm) are selected within the hypoxic area of the primary tumor. The distance between each spherical volume is 1.5 - 2 cm, and a high-dose radiotherapy of 12 Gy × 1F is delivered.
Drug: Tislelizumab, Carboplatin, Pemetrexed — For adenocarcinoma, pemetrexed (500 mg/m², day 1) + carboplatin (AUC 5, day 1) is used.
Drug: Tislelizumab, paclitaxel, Carboplatin — For NSCLC with pathological types other than adenocarcinoma, nab-paclitaxel (100 mg/m² on day 1 and day 8) + carboplatin (AUC 5, day 1) is used.

SUMMARY:
The aim of this clinical trial is to understand whether spatial fractionated radiotherapy (SFRT) in combination with tislelizumab and platinum-based doublet chemotherapy given concurrently as induction treatment is effective in treating initially unresectable stage Ⅲ non-small cell lung cancer (NSCLC). It will also explore the safety of this treatment modality. The main questions it aims to answer are:

Will spatial fractionated radiotherapy (SFRT) in combination with tislelizumab and platinum-based doublet chemotherapy given concurrently as induction treatment increase the surgical resection rate of patients with initially unresectable stage Ⅲ non-small cell lung cancer? What adverse reactions will patients experience when receiving spatial fractionated radiotherapy (SFRT) in combination with tislelizumab and platinum-based doublet chemotherapy given concurrently as induction treatment?

DETAILED DESCRIPTION:
Research Title: A Clinical Study on Induction Treatment with Spatial Fractionated Radiotherapy (SFRT) Concurrent with Tislelizumab Plus Platinum-based Doublet Chemotherapy for Initially Unresectable Stage III Non-small Cell Lung Cancer (NSCLC) Research Objective: To explore the efficacy and safety of induction treatment with spatial fractionated radiotherapy (SFRT) concurrent with tislelizumab plus platinum-based doublet chemotherapy for initially unresectable stage III non-small cell lung cancer (NSCLC).

Design Type: Interventional Study Research Subjects: Patients with non-small cell lung cancer diagnosed by pathological histology or cytology, staged as stage III (T3 - 4N1 - 2M0) according to the 8th edition of AJCC, defined as initially unresectable by the multidisciplinary team (MDT), without known EGFR and ALK mutations, aged ≥ 18 years old, with an ECOG PS score of 0 - 1.

Sample Size: 30 cases

ELIGIBILITY:
Inclusion Criteria:

* The patient has histologically or cytologically confirmed stage III non-small cell lung cancer (NSCLC) that is deemed unresectable after discussion in the multidisciplinary team (MDT), which is classified as T3-4N1-2M0 according to the 8th edition of the American Joint Committee on Cancer (AJCC).

Exclusion Criteria:

* Has participated in another clinical study using research products within the past 3 weeks.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Surgical resection rate | At the end of the surgery
  The percentage of patients who underwent surgical resection after induction treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Nanchang City, Jiangxi Province, Nanchang, Jiangxi, China